CLINICAL TRIAL: NCT01556607
Title: A Double-Blind, Randomized, 3 Period Crossover, Single Ascending Dose Study to Assess the Safety, and Tolerability of Inhaled MDT-637 in Subjects With Intermittent, or Mild-to-Moderate Persistent, Asthma
Brief Title: A Trial to Assess the Safety, Tolerability and Pharmacokinetics of MDT-637 in Subjects With Intermittent, or Mild-to-Moderate Persistent, Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicroDose Therapeutx, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDT-637-CP-103
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Drug Safety
Keywords: Respiratory Syncytial Virus Infection; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — VP-14637

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Experimental: MDT-637 (Active Comparator)
  Interventions: Drug: MDT-637
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDT-637 — Inhaled doses of MDT-637 over a 24 hour period at 3 visits
  Arms: Experimental: MDT-637
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MDT-637, when inhaled by subjects with Intermittent, or Mild-to-Moderate Persistent, Asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Documented clinical history and physician diagnosis of intermittent or mild or moderate persistent asthma for at least 6 months prior to screening OR subjects with historical record of Beta-agonist reversibility within previous 5 years
2. Subjects must demonstrate bronchial hyper-reactivity on methacholine challenge of PC20 less than 8mg/mL.
3. Visit 2 FEV1 (with no treatment change in the interim) must be within 12% of Visit 1 result
4. Males and/or females (if not surgically sterile or confirmed to be post menopausal) must agree to practice 2 barrier contraception methods until they are discharged from the study
5. Willing to give written informed consent
6. 18 to 50 years of age
7. BMI of 19-30 kg/m2
8. Non-smoker (for at least 90 days prior to screening) and willing to abstain from smoking during the course of the study
9. Good general health (excepting asthma) as determined by medical history, physical examination, ECG and clinical laboratory tests
10. Willing to abstain from alcohol, caffeine, and xanthine-containing beverages for 24 hours prior to dosing and for 24 hours after dosing.

Exclusion Criteria:

1. Uncontrolled, clinically significant disease which in the opinion of the Principal Investigator, Medical Monitor or Sponsor (MicroDose Therapeutx; MDTx) would place the subject at risk through study participation or would confound the assessment of the safety of MDT-637
2. Inability to perform acceptable and repeatable spirometry in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines
3. Abnormal FEV1, FVC, or FEV1/FVC (FEV1 and FVC < 75% of predicted and/or FEV1/FVC ratio < 0.7)
4. FEV1 variability > 12% between Visit 1 and Visit 2
5. Evidence of current or history of additional respiratory disease (other than asthma); for instance emphysema, chronic bronchitis or cystic fibrosis.
6. Upper respiratory tract infection within 6 weeks of Visit 1
7. Use of rescue albuterol or other short acting bronchodilator (SAB) more often than five times per week
8. History of significant nasal irritation from nasal inhalation of medication
9. History of malignancy
10. History of clinically significant alcohol or drug abuse
11. Positive drug screen for drugs of abuse
12. Positive test for HIV, Hepatitis B or Hepatitis C
13. Allergy to lactose, or lactose intolerance
14. Use of prescription medication (other than SAB and/or low dose inhaled corticosteroid e.g. fluticasone propionate 44 mcg BID or budesonide 100 mcg BID or equivalent) within 14 days of Visit 2 or over-the-counter preparations, including dietary and herbal supplements, within 5 days of Visit 2
15. Positive urine pregnancy test at Visit 1 or Visit 2 or visit 4
16. Abnormal QTc interval at Visit 1(> 450 msec in males or > 470 msec in females)
17. Significant blood donation (or testing) in previous 8 weeks
18. Use of any Investigational Product in previous 6 weeks (small molecule products) or previous 3 months (biologic products)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of escalating doses of MDT-637 when inhaled by subjects with Intermittent, or Mild-to-Moderate Persistent, Asthma. | Up to 61 days (including up to 42 days of screening period)
  Safety measurements include Clinical Laboratory Evaluations, Pulmonary Function Tests (Spirometry), ECG, Vital Signs, Physical Examination and Assessment of Adverse Events.

SECONDARY OUTCOMES:
Plasma pharmacokinetics for MDT-637 dry powder inhalation | Multiple plasma samples collected, upto 24 hr post last dose
  Plasma Samples will be measured to determine MDT-637 pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Purvee Shah, MD, Principal Investigator — West Coast Clinical Trials
Locations (1):
- West Coast Clinical Trials, Costa Mesa, California, United States

REFERENCES:
- See also: Development Program Information — http://mdtx.com/pipeline/proprietary-products/mdt-637/